CLINICAL TRIAL: NCT03357393
Title: Patient-controlled Sedation With Propofol Versus Combined Sedation During Bronchoscopy - a Randomized Controlled Trial
Brief Title: Patient-controlled Sedation With Propofol Versus Combined Sedation During Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lena Nilsson (Other)
Responsible Party: Sponsor-Investigator, Lena Nilsson, Principal Investigator, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRONSE
Record Dates: First submitted 2017-11-07; First posted 2017-11-29 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Sedation, Bronchoscopy
MeSH Terms: interventions — Midazolam; Propofol; Glycopyrrolate

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The bronchoscopist is blinded regarding given premedication for patients given PCS (two sedation arms).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midazolam and morphine-scopolamine (Active Comparator): Sedation during bronchoscopy with midazolam and morphine-scopolamine as premedication.
  Interventions: Drug: Midazolam; Drug: morphine-scopolamine
- PCS (propofol) with morphine-scopolamine (Experimental): Sedation during bronchoscopy with propofol using PCS and morphine-scopolamine as premedication
  Interventions: Drug: Propofol-Lipuro; Drug: morphine-scopolamine
- PCS (propofol) with glycopyrronium bromide (Experimental): Sedation during bronchoscopy with propofol using PCS and glycopyrronium bromide as premedication.
  Interventions: Drug: Propofol-Lipuro; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Midazolam — Midazolam is givenas sedation to the Control arm.
  Arms: Midazolam and morphine-scopolamine
Drug: Propofol-Lipuro — Propofol is given as sedation to both intervention arms.
  Arms: PCS (propofol) with glycopyrronium bromide; PCS (propofol) with morphine-scopolamine
Drug: morphine-scopolamine — Given as premedication for the Control arm and one of the interventions arms.
  Arms: Midazolam and morphine-scopolamine; PCS (propofol) with morphine-scopolamine
Drug: Glycopyrrolate — Given as premedication for one of the intervention arms..
  Arms: PCS (propofol) with glycopyrronium bromide

SUMMARY:
bronchoscopy - a randomized controlled trial" (EudraCT number: 2015-005274-38, protocol number: "BRONSE") is a phase IV single centre prospective randomized controlled trial with parallel groups. A total of 150 adult outpatients undergo diagnostic bronchoscopy during sedation and are randomized into three sedation arms (1:1:1); sedation with midazolam and morphine-scopolamine as premedication (clinical routine), sedation with propofol using PCS and morphine-scopolamine as premedication, and sedation with propofol using PCS and glycopyrronium bromide as premedication. The study is partially blinded, the bronchoscopist is blinded regarding given premedication for patients given PCS (two sedation arms). The hypothesis is that PCS increase the amount of patients ready for discharge, and further that patient characteristics affect the amount of propofol administered. The endpoints are primarily the amount of patients ready for discharge within 2 hours and secondary assessment of patient recovery and satisfaction as well as bronchoscopist evaluation and doses of administrated drugs. Finally safety variables are collected such as vital signs and interventions performed to maintain cardiovascular and respiratory stability.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Planned bronchoscopic procedure with sedation in an outpatient setting
* The patient have after receiving information about the study given his/her signed informed consent to participate.
* Women of childbearing potential only if use of effective contraceptive.

Exclusion Criteria:

* Positive pregnancy test S-β-HCG.
* Known/suspected allergy or contraindication* to any medication within the study.
* Functional disability in both hands which affect the possibility to operate the PCS device.
* Cognitive impairment, unwillingness or language difficulties resulting in difficulty to understand the meaning of participation in the study or to operate the PCS device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Median (Full Range); unit: years] | 70 [33 to 83] | 69 [25 to 86] | 68 [25 to 89] | 69 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 28 | 72
  Male | 28 | 28 | 22 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Discharge Assessment Using PADSS After 2 Hours Number of Patients Reaching PADSS Score 10 After 2 Hours
Description: Post Anaesthetic Discharge Scoring System (PADSS).A measurement of the PADSS score is done by pulmonary nurse every 15 min after bronchoscopy is finished (when bronchoscope is removed) for 2 hours. The PADSS is used to clinically assess if the patient is ready to be discharged after anaesthesia/sedation and consist of five criteria: vital signs, ambulation, nausea and/or vomiting, pain and surgical bleeding. Each criterion is given a score ranging from 0 to 2. Only patients who achieve a total score of 10 are considered ready for discharge after 2 hours.
Time Frame: 2 hours after bronchoscopy is finished
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
Participants | 19 | 30 | 45

2. Secondary Outcome: Assessment of Self-rated Patient Questionaries' Using S-PSR
Description: Post-discharge Surgical Recovery Scale (S-PSR) The modified Swedish version S-PSR is based on the "Post-discharge Surgical Recovery Scale" and is a 14-item questionnaire to assess the recovery post-discharge regarding the patients' health status and activity (see further appendix 2). Each item is rated using a semantic differential scale and the total sum is multiplied by 100. The possible range is 10-100, with higher score indicating a more favourable postoperative recovery.
Time Frame: The assessment is done by the patient at home (or at ward if pro-longed hospital stay is necessary) in the evening on the day of bronchoscopy. It takes approximately 2 minutes to complete the questionnaire.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 55 [36 to 77] | 56 [43 to 73] | 54 [41 to 100]

3. Secondary Outcome: Quality of Recovery (QoR-23)
Description: Modified version of Quality of Recovery (QoR-23) Minimum value 23. Maximum value 115. A higher score indicate a better quality of recovery.
  The questionnaire "Quality of Recovery" (QoR-23) is a 23 item questionnaire to assess recovery after day surgery regarding the patients' emotional state, physical comfort and physical independence (see further appendix 4). Each item is rated on a five-point scale (1-5) and the scores are summed.
Time Frame: The assessment is done by the patient at home (or at ward if pro-longed hospital stay is necessary) in the morning the day after bronchoscopy. It takes less than 1 minute to complete the assessment.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
score on a scale | 100 [61 to 112] | 102 [60 to 115] | 100 [63 to 115]

4. Secondary Outcome: Patients' Satisfaction Using a Likert-type Scale
Description: overall satisfaction with the procedure using the Likert-type scale (1. Very dissatisfied, 2. Dissatisfied, 3. Neither satisfied nor dissatisfied, 4. Satisfied, 5. Very satisfied). The patient may comment any cause which made the satisfaction score high or low and if the patient would like to receive the same method of sedation during a future bronchoscopy.
Time Frame: After patient has recovered after bronchoscopy and before discharge home, estimated period of time 0-24 hours.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 5 [2 to 5] | 5 [4 to 5] | 5 [4 to 5]

5. Secondary Outcome: Bronchoscopist Evaluation Using a Likert-type Scale
Description: the bronchoscopist assess their perception of cough, bronchial secretion respectively circumstances for a smooth performance of the bronchoscopy of procedure using the Likert-type scale (1. Very dissatisfied, 2. Dissatisfied, 3. Neither satisfied nor dissatisfied, 4. Satisfied, 5. Very satisfied).
Time Frame: Directly after completion of the procedure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 5 [2 to 5] | 4 [1 to 5] | 4 [2 to 5]

6. Other Pre Specified Outcome: Level of Sedation Using the Observer's Assessment of Alertness/Sedation (OAA/S) Scale
Description: Level of sedation is assessed every 5th minute during the procedure by the nurse anaesthetist using The Observer's Assessment of Alertness/Sedation (OAA/S) scale whereby a higher score represent a lighter sedation. Below is the scale descriped, Observation/score:
  Responds readily to name spoken in normal tone/5 Lethargic response to name spoken in normal tone/4 Responds only after name is called loudly and/or repeatedly/3 Responds only after mild prodding or shaking/2 Does not respond to mild prodding or shaking/1
Time Frame: Assessement are done every 5th minute from procedure start until end of procedure (extraction of bronchoscope), estimated period of time 0-60 minutes.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 3 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]

7. Other Pre Specified Outcome: Number of Participants With Interventions Performed
Description: Number of participants with interventions performed to maintain cardiovascular (if atropine or ephidrine has been given) and respiratory stability (if assisted ventilation, chin lift or painful stimulation has been performed). Assesed every five minutes during the procedure.
Time Frame: From procedure start until end of procedure (extraction of bronchoscope), estimated period of time 0-60 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
Number analyzed (Participants) | 50 | 50 | 50
Participants | 1 | 4 | 3

8. Other Pre Specified Outcome: Arterial Oxygen Saturation (SpO2)
Time Frame: Every five minutes during the procedure (from procedure start until end of procedure (extraction of bronchoscope), , estimated period of time 0-60 minutes, and thereafter after the procedure every 15 minutes until PADSS score ≥9 or maximum 4 hours.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Respiratory Rate Per Minute (RR)
Time Frame: as for outcome 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Non-invasive Blood Pressure (mmHg)
Time Frame: as for outcome 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Heart Rate (Beats Per Minute, HR).
Time Frame: as for outcome 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From start preparation for bronchospcpy (first drug given) to completing the questionnary QoR-23 on the day after procedure
Description: In the incident report the following grading is used to rate the severity of an incidence:
  * Mild = aware of the symptoms but they are tolerable
  * Moderate = symptoms partially affect daily activities
  * Severe = symptoms significantly affect daily activities
  The investigator assesses the relationship between the incidence and the study, as defined:
  • Likely = good reasons and sufficient documentation to suspect caus
Arm/Group | Midazolam and Morphine-scopolamine | PCS (Propofol) With Morphine-scopolamine | PCS (Propofol) With Glycopyrronium Bromide
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 3/50 | 6/50 | 2/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam and Morphine-scopolamine (N=50) | PCS (Propofol) With Morphine-scopolamine (N=50) | PCS (Propofol) With Glycopyrronium Bromide (N=50)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Severe short bradycardia during sedaation. Required pharmacological treatment
Overnight admission (General disorders) | 3 (3) | 0 (0) | 0 (0) — Unplanned overnight admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam and Morphine-scopolamine (N=50) | PCS (Propofol) With Morphine-scopolamine (N=50) | PCS (Propofol) With Glycopyrronium Bromide (N=50)
Dizzyness, confusion (General disorders) | 3 (3) | 6 (6) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03357393/Prot_SAP_000.pdf